CLINICAL TRIAL: NCT03538717
Title: Retrospective Analysis of Clinical Factors Associated With Greater Benefit of Axitinib in Metastatic Renal Cancer (AXILONG Study)
Brief Title: "Retrospective Study to Identify Clinical Factors Related to a High Benefit of Axitinib in mRCC"
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A4061089; AXILONG (Other: Alias Study Number)
Record Dates: First submitted 2018-01-19; First posted 2018-05-29 (Actual); Results first posted 2020-03-13 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Carcinoma, Renal Cell
Keywords: Axitinib,; Renal Carcinoma,; Long responders
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Retrospective study to collect data from Patients with advanced/metastatic renal cell carcinoma previously treated with Axitinib under standard clinical practice, to describe the clinical profile of the patients with a long response to Axitinib and to try to identify clinical factors which could be related with the long response to Axitinib, through the comparison between long responder patients and a group of refractory patients

DETAILED DESCRIPTION:
To describe the clinical profile of patients with a long response to Axitinib and to identify clinical factors which could be related with the long response to Axitinib, through the comparison between long responder patients and a group of refractory patients.

For this study are defined as "long responder", those patients who has a Progression Free Survival (PFS) of at least 9 months since the initiation of Axitinib treatment, and "refractory patients" those who have Progression Disease (PD) in the first response assessment since the initiation of Axitinib treatment (estimated PFS ≤3 months]

Secondary Objectives

* To describe the efficacy of Axitinib treatment in the long responders group, and in relation with the treatment received before Axitinib, in terms of PFS, ORR, CB, OS, TTP ...
* To describe the tolerability and drug management of Axitinib in this population.
* To describe treatment received after Axitinib in this population.

Study procedures:

For the recruitment, the Investigator should review the inclusion / exclusion criteria. In case of patients alive at the moment of the inclusion, the investigator will require them to sign the IC.

With the data available in the medical records, the information requested will be recorded in the electronic data collection tool.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years

  * Patients with advanced or metastatic renal cell carcinoma, histologically confirmed, with at least one radiological response assessment
  * Patients who had received Axitinib treatment in second or further line with a PFS ≥9 months or DP (disease progression) at the first tumor assessment.
  * For the patients alive at the moment of the inclusion, patients must have a signed informed consent document

Exclusion Criteria:

* Axitinib received out of the approved indication Patients who do not meet any of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Age ≥ 18 years
  * Patients with advanced or metastatic renal cell carcinoma, histologically confirmed, with at least one radiological response assessment
  * Patients who had received Axitinib treatment in second or further line with a PFS ≥9 months or DP (disease progression) at the first tumor assessment.
  * For the patients alive at the moment of the inclusion, patients must have a signed informed consent document
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (40):
- Spain (40):
  - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Parc Taulí, Sabadell, Barcelona
  - Hospital Sant Pau i Santa Tecla, Tarragona, Barcelona
  - Hospital Universitario Mutua Terrassa, Terrassa, Barcelona
  - Complejo Hospitalario la Mancha Centro, Alcázar de San Juan, Ciudad REAL
  - Hospital Universitario Principe de Asturias, Alcalá de Henares, Madrid
  - Hospital Universitario Fundacion Alcorcón, Alcorcón, Madrid
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Universitario Rey Juan carlos, Móstoles, Madrid
  - Hospital Infanta Cristina, Parla, Madrid
  - Hospital Universitario Infanta Sofía, San Sebatián de Los Reyes, Madrid
  - Hospital Universitario Son Espases, Palma de Mallorca, Mallorca
  - HU de Navarra, Pamplona, Pamplona, Navarre
  - Hospital Universitario de Canarias, La Cuesta, Santa Cruz de Tenerife, Tenerife
  - Hospital Universitario Nuestra Señora de la Candelaria, Tenerife, Santa Cruz de Tenerife, Tenerife
  - Hospita General Nuestra Señora del Prado, Talavera de la Reina, Toledo
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebrón, Barcelona
  - HU Clinic i Provincial, Barcelona
  - Hospital Universitario Sant Pau i Santa Creu, Barcelona
  - Hospital General Universitario de Ciudad Real, Ciudad Real
  - Hospital Reina Sofía, Córdoba
  - Complejo Hospitalario de Jaén, Jaén
  - HU De León, León
  - Hospital Universitario Lucus Augusti (HULA_ Lugo), Lugo
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Fundación Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Centro Integral Oncológico Clara Campal, Madrid
  - Complejo Hospitalario Universitario de Ourense CHUOU, Ourense
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Santiago de Compostela, Santiago de Compostela
  - Hospita Virgen de la Salud de Toledo, Toledo
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Universitario de Vigo- Hospital Álvaro Cunqueiro, Vigo
  - H. Universitario Miguel Servet, Zaragoza, Zaragoza
  - Hospital Clínico Uiversitario Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A4061089

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data was collected and observed retrospectively for approximately 1 year, of metastatic renal cell carcinoma (mRCC) participants who received axitinib in the daily clinical practice as second and later lines prior to inclusion in study and met inclusion/exclusion criteria.
Groups:
- Axitinib (INLYTA): Participants with advanced or mRCC who had been treated with axitinib before inclusion in this study, under standard clinical practice as a second-line treatment or further line as per its summary of product characteristics and had a progression free survival of at least 9 months (long responders) or had disease progression as best response to this treatment (refractory). During this study, data for these participants was collected and observed retrospectively, for approximately 1 year.
Period: Overall Study
Arm/Group | Axitinib (INLYTA)
Started | 157
Completed | 157
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all evaluable participants, i.e. all participants who met all the inclusion criteria and none of the exclusion criteria and had received at least 1 dose of axitinib prior to inclusion in the study.
Arm/Group | Axitinib (INLYTA)
Number analyzed (Participants) | 157
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: 1 participant had an erroneous birth date data, hence data was not included for that participant.
  Years
    number analyzed (Participants) | 156
    (all) | 59.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 120
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Age Less Than or Equal to (<=) 65 Years and Greater Than (>) 65 Years at Initiation of Axitinib Treatment: Long Responders Versus Refractory Participants
Time Frame: At initiation of axitinib treatment, within axitinib therapy of maximum 5.4 years approximately (from the data collected and observed retrospectively during 1 year)
Population: FAS included all evaluable participants, i.e. all participants who met all the inclusion criteria and none of the exclusion criteria and have received at least 1 dose of axitinib prior to inclusion in the study. Here, "Overall Number of Participants" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Long Responders to Axitinib: Participants with advanced or mRCC who had been treated with axitinib, under standard clinical practice as a second-line treatment or further line as per its summary of product characteristics and had a progression-free survival of at least 9 months with axitinib treatment. During this study, data for these participants was collected and observed, retrospectively for approximately 1 year.
- Axitinib Refractory Participants: Participants with advanced or mRCC who had been treated with axitinib, under standard clinical practice as a second-line treatment or further line as per its summary of product characteristics and had disease progression as best response to this treatment and had disease progression at the first assessment after the initiation of treatment (estimated PFS was <=3 months). During this study, data for these participants was collected and observed, retrospectively for approximately 1 year.
Arm/Group | Long Responders to Axitinib | Axitinib Refractory Participants
Number analyzed (Participants) | 91 | 65
Participants
  <= 65 years | 58 | 50
  > 65 years | 33 | 15
Statistical Analysis 1: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; Statistics analysis (P value) was performed compositely for all the categories reported; Test type: Superiority; p = 0.113, Chi-squared

2. Primary Outcome: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status Before First Line Treatment Initiation: Long Responders Versus Refractory Participants
Description: ECOG: participant's performance status was measured on a 6-point scale: 0= fully active/able to carry on all pre-disease activities without restriction; 1= restricted in physically strenuous activity but ambulatory and able to carry out work of a light and sedentary nature; 2= ambulatory and capable of all self-care, but unable to carry out any work activities, up and about more than 50 percent (%) of waking hours; 3= capable of only limited self-care, confined to bed/chair >50% of waking hours; 4= completely disabled, cannot carry on any self-care, totally confined to bed/chair: 5= dead. In this outcome measure, data for ECOG status (0, 1, >=2: before first line treatment initiation), was compared between long responders and refractory participants.
Time Frame: Prior to first dose of first line treatment, within first line therapy of maximum 6.6 years approximately (from the data collected and observed retrospectively during 1 year)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Long Responders to Axitinib | Axitinib Refractory Participants
Number analyzed (Participants) | 75 | 53
Participants
  ECOG: 0 | 49 | 28
  ECOG: 1 | 23 | 24
  ECOG: >=2 | 3 | 1
Statistical Analysis 1: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; Statistics analysis (P value) was performed compositely for all the categories reported; Test type: Superiority; p = 0.228, Fisher Exact

3. Primary Outcome: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status at Initiation of Axitinib Treatment: Long Responders Versus Refractory Participants
Description: ECOG: participant's performance status was measured on a 6-point scale: 0= fully active/able to carry on all pre-disease activities without restriction; 1= restricted in physically strenuous activity but ambulatory and able to carry out work of a light and sedentary nature; 2= ambulatory and capable of all self-care, but unable to carry out any work activities, up and about more than 50 percent (%) of waking hours; 3= capable of only limited self-care, confined to bed/chair >50% of waking hours; 4= completely disabled, cannot carry on any self-care, totally confined to bed/chair: 5= dead. In this outcome measure, data for ECOG status (0, 1, >=2: at initiation of axitinib), was compared between long responders and refractory participants.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Long Responders to Axitinib | Axitinib Refractory Participants
Number analyzed (Participants) | 80 | 52
Participants
  ECOG: 0 | 34 | 10
  ECOG: 1 | 39 | 34
  ECOG: >=2 | 7 | 8
Statistical Analysis 1: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; Statistics analysis (P value) was performed compositely for all the categories reported; Test type: Superiority; p = 0.020, Chi-squared

4. Primary Outcome: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status on Axitinib Discontinuation: Long Responders Versus Refractory Participants
Description: ECOG: participant's performance status was measured on a 6-point scale: 0= fully active/able to carry on all pre-disease activities without restriction; 1= restricted in physically strenuous activity but ambulatory and able to carry out work of a light and sedentary nature; 2= ambulatory and capable of all self-care, but unable to carry out any work activities, up and about more than 50 percent (%) of waking hours; 3= capable of only limited self-care, confined to bed/chair >50% of waking hours; 4= completely disabled, cannot carry on any self-care, totally confined to bed/chair: 5= dead. In this outcome measure, data for ECOG status (0, 1, >=2: on axitinib discontinuation), was compared between long responders and refractory participants.
Time Frame: On discontinuation of axitinib treatment, within axitinib therapy of maximum 5.4 years approximately (from the data collected and observed retrospectively during 1 year)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Long Responders to Axitinib | Axitinib Refractory Participants
Number analyzed (Participants) | 61 | 53
Participants
  ECOG: 0 | 16 | 9
  ECOG: 1 | 32 | 24
  ECOG: >=2 | 13 | 20
Statistical Analysis 1: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; Statistics analysis (P value) was performed compositely for all the categories reported; Test type: Superiority; p = 0.138, Chi-squared

5. Primary Outcome: Number of Participants With 1 or More Different Treatment Lines Before Axitinib Treatment Initiation: Long Responders Versus Refractory Participants
Time Frame: Prior to first dose of axitinib treatment, within axitinib therapy of maximum 5.4 years approximately (from the data collected and observed retrospectively during 1 year)
Population: FAS included all evaluable participants, i.e. all participants who met all the inclusion criteria and none of the exclusion criteria and have received at least 1 dose of axitinib prior to inclusion in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Long Responders to Axitinib | Axitinib Refractory Participants
Number analyzed (Participants) | 91 | 66
Participants
  1 Treatment Line | 58 | 48
  2 Treatment Lines | 18 | 10
  >=3 Treatment Lines | 15 | 8
Statistical Analysis 1: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; Statistics analysis (P value) was performed compositely for all the categories reported; Test type: Superiority; p = 0.524, Chi-squared

6. Primary Outcome: Number of Participants With Nephrectomy Procedure Status Before Axitinib Treatment Initiation: Long Responders Versus Refractory Participants
Description: Nephrectomy is a surgical removal of kidney. Data for participants was categorized as yes and no to depict their nephrectomy status before axitinib treatment initiation and comparison was done between long responders and refractory participants.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Long Responders to Axitinib | Axitinib Refractory Participants
Number analyzed (Participants) | 91 | 66
Participants
  Yes | 85 | 58
  No | 6 | 8
Statistical Analysis 1: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; Statistics analysis (P value) was performed compositely for all the categories reported; Test type: Superiority; p = 0.265, Chi-squared

7. Primary Outcome: Number of Participants With Memorial Sloan Kettering Cancer Center (MSKCC) Risk Group Before First Line Treatment Initiation: Long Responders Versus Refractory Participants
Description: MSKCC risk system stratifies participants with mRCC into poor, intermediate and favorable risk groups based on number of adverse clinical and laboratory parameters present. Favorable-risk group: participants had no poor prognostic factors. Intermediate-risk group: participants had 1 or 2 adverse prognostic factors. Poor-risk group: participants had more than 2 poor prognostic factors. Poor prognostic factors included a Karnofsky performance status (KPS) of less than (<) 80 (KPS score quantify participant's general well-being and activities of daily life, based on their functional impairment. KPS score ranges between 0= death to 100= no evidence of disease; higher score means higher ability to perform daily tasks), time from diagnosis to treatment for more than 12 months, serum lactate dehydrogenase (LDH) >1.5*upper limit of normal (ULN), corrected serum calcium level >10.0 milligram per deciliter (mg/dL) and hemoglobin < lower limit of normal (LLN).
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Long Responders to Axitinib | Axitinib Refractory Participants
Number analyzed (Participants) | 47 | 44
Participants
  Favorable risk group | 15 | 7
  Intermediate risk group | 25 | 21
  Poor risk group | 7 | 16
Statistical Analysis 1: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; Statistics analysis (P value) was performed compositely for all the categories reported; Test type: Superiority; p = 0.035, Chi-squared

8. Primary Outcome: Number of Participants With Memorial Sloan Kettering Cancer Center (MSKCC) Risk Group at Initiation of Axitinib Treatment: Long Responders Versus Refractory Participants
Description: MSKCC risk system stratifies participants with mRCC into poor, intermediate and favorable risk groups based on number of adverse clinical and laboratory parameters present. Favorable-risk group: participants had no poor prognostic factors. Intermediate-risk group: participants had 1 or 2 adverse prognostic factors. Poor-risk group: participants had more than 2 poor prognostic factors. Poor prognostic factors included a KPS of <80 (KPS score quantify participant's general well-being and activities of daily life, based on their functional impairment. KPS score ranges between 0= death to 100= no evidence of disease; higher score means higher ability to perform daily tasks), time from diagnosis to treatment for more than 12 months, serum LDH >1.5*ULN, corrected serum calcium level >10.0 mg/dL and hemoglobin < LLN.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Long Responders to Axitinib | Axitinib Refractory Participants
Number analyzed (Participants) | 65 | 46
Participants
  Favorable risk group | 13 | 7
  Intermediate risk group | 28 | 13
  Poor risk group | 24 | 26
Statistical Analysis 1: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; Statistics analysis (P value) was performed compositely for all the categories reported; Test type: Superiority; p = 0.123, Chi-squared

9. Primary Outcome: Number of Participants With Memorial Sloan Kettering Cancer Center (MSKCC) Risk Group on Discontinuation of Axitinib Treatment: Long Responders Versus Refractory Participants
Description: as for outcome 8
Time Frame: On discontinuation of axitinib treatment, within axitinib therapy during treatment of maximum 5.4 years, approximately (from the data collected and observed retrospectively during 1 year)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Long Responders to Axitinib | Axitinib Refractory Participants
Number analyzed (Participants) | 49 | 44
Participants
  Favorable risk group | 10 | 6
  Intermediate risk group | 26 | 20
  Poor risk group | 13 | 18
Statistical Analysis 1: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; Statistics analysis (P value) was performed compositely for all the categories reported; Test type: Superiority; p = 0.327, Chi-squared

10. Primary Outcome: Number of Participants With International Metastatic Database Consortium (IMDC) Risk Group at Initiation of Axitinib Treatment: Long Responders Versus Refractory Participants
Description: IMDC risk group stratifies participants with mRCC into poor, intermediate and favorable risk groups based on number of adverse clinical and laboratory parameters present. Favorable-risk group: participants had no poor prognostic factors. Intermediate-risk group: participants had 1 or 2 poor prognostic factors. Poor-risk group: participants had 3 to 6 poor prognostic factors. Poor prognostic factors included KPS score of <80 at the initiation of treatment, time from diagnosis to metastasis treatment of <12 months, anemia, hypercalcemia (corrected calcium >10 mg/dL), neutrophilia and thrombocythemia. In this outcome measure, IMDC risk group (favorable, intermediate, poor: at initiation of axitinib) was compared between long responders and refractory participants.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Long Responders to Axitinib | Axitinib Refractory Participants
Number analyzed (Participants) | 65 | 43
Participants
  Favorable risk group | 6 | 4
  Intermediate risk group | 37 | 19
  Poor risk group | 22 | 20
Statistical Analysis 1: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; Statistics analysis (P value) was performed compositely for all the categories reported; Test type: Superiority; p = 0.419, Chi-squared

11. Primary Outcome: Number of Participants With International Metastatic Database Consortium (IMDC) Risk Group on Discontinuation of Axitinib Treatment: Long Responders Versus Refractory Participants
Description: IMDC risk group stratifies participants with mRCC into poor, intermediate and favorable risk groups based on number of adverse clinical and laboratory parameters present. Favorable-risk group: participants had no poor prognostic factors. Intermediate-risk group: participants had 1 or 2 poor prognostic factors. Poor-risk group: participants had 3 to 6 poor prognostic factors. Poor prognostic factors included KPS score of <80 at the initiation of treatment, time from diagnosis to metastasis treatment of <12 months, anemia, hypercalcemia (corrected calcium >10 mg/dL), neutrophilia and thrombocythemia. In this outcome measure, IMDC risk group (favorable, intermediate, poor: on discontinuation of axitinib) was compared between long responders and refractory participants.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Long Responders to Axitinib | Axitinib Refractory Participants
Number analyzed (Participants) | 51 | 44
Participants
  Favorable risk group | 4 | 5
  Intermediate risk group | 33 | 15
  Poor risk group | 14 | 24
Statistical Analysis 1: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; Statistics analysis (P value) was performed compositely for all the categories reported; Test type: Superiority; p = 0.010, Fisher Exact

12. Primary Outcome: Number of Participants With Different Type of Renal Cells Before Axitinib Treatment Initiation: Long Responders Versus Refractory Participants
Description: In this outcome measure, data for participants who had renal cells with different type of histology as 100% clear cells, 100% non-clear cells, majority component of clear cells and majority component of non-clear cells was compared between long responders and refractory participants.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Long Responders to Axitinib | Axitinib Refractory Participants
Number analyzed (Participants) | 91 | 65
Participants
  100% clear cells | 72 | 48
  100% non-clear cells | 8 | 8
  Majority component of clear cells | 7 | 7
  Majority component of non-clear cells | 4 | 2
Statistical Analysis 1: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; 100% clear cells; Test type: Superiority; p = 0.446, Chi-squared
Statistical Analysis 2: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; 100% non-clear cells; Test type: Superiority; p = 0.596, Chi-squared
Statistical Analysis 3: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; Majority component of clear cells; Test type: Superiority; p = 0.578, Chi-squared
Statistical Analysis 4: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; Majority component of non-clear cells; Test type: Superiority; p = 0.706, Fisher Exact

13. Primary Outcome: Number of Participants With Duration of First Line Treatment With Tyrosine Kinase Inhibitor (TKI) Before Axitinib Treatment Initiation: Long Responders Versus Refractory Participants
Description: Duration of first line treatment with TKI was stratified into 0-3 months, 3-6 months, 6-9 months, 9-12 months and >12 months and compared between long responders and refractory participants.
Time Frame: First dose of first line treatment, within first line therapy of maximum 6.6 years approximately (from the data collected and observed retrospectively during 1 year)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Long Responders to Axitinib | Axitinib Refractory Participants
Number analyzed (Participants) | 88 | 62
Participants
  0-3 months | 6 | 6
  3-6 months | 7 | 13
  6-9 months | 6 | 7
  9-12 months | 13 | 9
  >12 months | 56 | 27
Statistical Analysis 1: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; Statistics analysis (P value) was performed compositely for all the categories reported; Test type: Superiority; p = 0.074, Chi-squared

14. Primary Outcome: Number of Participants With Best Response to First Line Treatment With Tyrosine Kinase Inhibitor (TKI) Before Axitinib Treatment Initiation: Long Responders Versus Refractory Participants
Description: In this outcome measure, data for participants with their best response as complete response (CR) and partial response (PR), stable disease (SD) or progressive-disease (PD) to the first line treatment with TKI, was compared between long responders and refractory participants. As per response evaluation criteria in solid tumors (RECIST) 1.1 criteria: CR = disappearance of all target lesions. PR = greater than equal to (>=) 30% decrease in sum of target lesions taking as reference baseline sum diameters. PD: >= 20% increase in sum of diameters of target lesions, taking as a reference smallest sum on treatment, the sum must also demonstrate an absolute increase of at least 5 millimeter (mm), or the appearance of >=1 new lesions. SD =neither shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters during treatment.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Long Responders to Axitinib | Axitinib Refractory Participants
Number analyzed (Participants) | 89 | 59
Participants
  CR+PR | 53 | 24
  SD | 26 | 24
  PD | 10 | 11
Statistical Analysis 1: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; Statistics analysis (P value) was performed compositely for all the categories reported; Test type: Superiority; p = 0.070, Chi-squared

15. Primary Outcome: Number of Participants With 1 or More Metastatic Locations at Diagnosis of Advance or Metastatic Renal Cell Carcinoma Before First Line Treatment Initiation: Long Responders Versus Refractory Participants
Time Frame: At diagnosis of advance or mRCC prior to first dose of first line treatment, within first line therapy of maximum 6.6 years approximately (from the data collected and observed retrospectively during 1 year)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Long Responders to Axitinib | Axitinib Refractory Participants
Number analyzed (Participants) | 91 | 66
Participants
  1 | 56 | 29
  2 | 23 | 23
  >=3 | 12 | 14
Statistical Analysis 1: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; Statistics analysis (P value) was performed compositely for all the categories reported; Test type: Superiority; p = 0.091, Chi-squared

16. Primary Outcome: Number of Participants With Different Metastatic Sites Locations at Diagnosis of Advance or Metastatic Renal Cell Carcinoma Before Axitinib Treatment Initiation: Long Responders Versus Refractory Participants
Description: In this outcome measure, data for participants with different metastatic sites as lymph nodes, central nervous system (CNS), hepatic, pulmonary, bone and another site of metastasis at diagnosis of advance or mRCC before axitinib treatment initiation, was compared between long responders and refractory participants.
Time Frame: as for outcome 15
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Long Responders to Axitinib | Axitinib Refractory Participants
Number analyzed (Participants) | 91 | 66
Participants
  Lymph nodes | 28 | 31
  CNS | 3 | 2
  Hepatic | 9 | 16
  Pulmonary | 56 | 35
  Bone | 12 | 19
  Another site of metastasis | 35 | 16
Statistical Analysis 1: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; Lymph nodes; Test type: Superiority; p = 0.046, Chi-squared
Statistical Analysis 2: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; CNS; Test type: Superiority; p > 0.999, Fisher Exact
Statistical Analysis 3: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; Hepatic; Test type: Superiority; p = 0.026, Chi-squared
Statistical Analysis 4: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; Pulmonary; Test type: Superiority; p = 0.327, Chi-squared
Statistical Analysis 5: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; Bone; Test type: Superiority; p = 0.024, Chi-squared
Statistical Analysis 6: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; Another site of metastasis; Test type: Superiority; p = 0.045, Chi-squared

17. Primary Outcome: Number of Participants With Laboratory Parameters at Initiation of First Line Treatment: Long Responders Versus Refractory Participants
Description: In this outcome measure, data for different laboratory parameters at initiation of first line treatment: LDH level >1.5*ULN, haemoglobin (Hgb) levels <=LLN, corrected Ca levels >10 mg/dL, neutrophil levels >ULN, platelet levels >ULN and neutrophil-to-lymphocyte ratio of <=3 was compared between long responders and refractory participants.
Time Frame: At initiation of first line treatment, within first line therapy of maximum 6.6 years approximately (from the data collected and observed retrospectively during 1 year)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Long Responders to Axitinib | Axitinib Refractory Participants
Number analyzed (Participants) | 91 | 66
Participants
  LDH level >1.5*ULN: number analyzed (Participants) | 66 | 51
  LDH level >1.5*ULN: Yes | 6 | 7
  LDH level >1.5*ULN: No | 60 | 44
  Hgb levels <=LLN: number analyzed (Participants) | 80 | 61
  Hgb levels <=LLN: Yes | 10 | 27
  Hgb levels <=LLN: No | 70 | 34
  Corrected Ca levels >10 mg/dL: number analyzed (Participants) | 55 | 50
  Corrected Ca levels >10 mg/dL: Yes | 4 | 7
  Corrected Ca levels >10 mg/dL: No | 51 | 43
  Neutrophil levels >ULN: number analyzed (Participants) | 79 | 58
  Neutrophil levels >ULN: Yes | 12 | 8
  Neutrophil levels >ULN: No | 67 | 50
  Platelet levels >ULN: number analyzed (Participants) | 80 | 59
  Platelet levels >ULN: Yes | 9 | 8
  Platelet levels >ULN: No | 71 | 51
  Neutrophil-to-lymphocyte ratio <=3: number analyzed (Participants) | 71 | 52
  Neutrophil-to-lymphocyte ratio <=3: Yes | 22 | 23
  Neutrophil-to-lymphocyte ratio <=3: No | 49 | 29
Statistical Analysis 1: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; LDH level >1.5*ULN; Test type: Superiority; p = 0.555, Chi-squared
Statistical Analysis 2: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; Hgb levels <=LLN; Test type: Superiority; p < 0.001, Chi-squared
Statistical Analysis 3: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; Corrected Ca levels >10 mg/dL; Test type: Superiority; p = 0.344, Chi-squared
Statistical Analysis 4: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; Neutrophil levels >ULN; Test type: Superiority; p > 0.999, Chi-squared
Statistical Analysis 5: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; Platelet levels >ULN; Test type: Superiority; p = 0.795, Chi-squared
Statistical Analysis 6: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; Neutrophil-to-lymphocyte ratio <=3; Test type: Superiority; p = 0.184, Chi-squared

18. Primary Outcome: Number of Participants With Smoking Habits at Initiation of First Line Treatment: Long Responders Versus Refractory Participants
Description: In this outcome measure, data for smoking habit of participants was compared between long responders and refractory participants.
Time Frame: as for outcome 17
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Long Responders to Axitinib | Axitinib Refractory Participants
Number analyzed (Participants) | 85 | 66
Participants
  Smoker | 34 | 26
  Non-smoker | 13 | 17
  Ex-smoker | 38 | 23
Statistical Analysis 1: Comparison: Long Responders to Axitinib vs Axitinib Refractory Participants; Statistics analysis (P value) was performed compositely for all the categories reported; Test type: Superiority; p = 0.235, Chi-squared

19. Secondary Outcome: Progression-free Survival (PFS) to Axitinib Treatment in Group of Long Responders
Description: PFS was defined as the time from the start of axitinib treatment to disease progression or death by any cause. If there was no progression or death, the case was censored as PFS at date of latest follow-up. PD: >= 20% increase in sum of diameters of target lesions, taking as a reference smallest sum on treatment, the sum must also demonstrate an absolute increase of at least 5 mm, or the appearance of >=1 new lesions.
Time Frame: Day 1 of axitinib dose to disease progression or death due to any cause or date of latest follow-up in case of censored up to a maximum axitinib therapy of 5.4 years, approximately (from the data collected and observed retrospectively during 1 year)
Population: FAS included all evaluable participants, i.e. all participants who met all the inclusion criteria and none of the exclusion criteria and have received at least 1 dose of axitinib prior to inclusion in the study. This outcome measure as per protocol was intended to be analyzed only in long responders group.
Measure: Median (Standard Error); unit: months
Arm/Group | Long Responders to Axitinib
Number analyzed (Participants) | 91
months | 18.136 (2.230)

20. Secondary Outcome: Time to Progression (TTP) to Axitinib Treatment in Group of Long Responders
Description: TTP was defined as the time from the start of axitinib treatment to date of disease progression. If there was no progression, the case was censored as TTP at latest follow-up. As per RECIST 1.1, PD: >= 20% increase in sum of diameters of target lesions, taking as a reference smallest sum on treatment, the sum must also demonstrate an absolute increase of at least 5 mm, or the appearance of >=1 new lesions.
Time Frame: Day 1 of axitinib dose to disease progression or date of latest follow-up in case of censored up to a maximum (max.)axitinib therapy duration of 5.4 years(yrs.)approximately(approx.)(from the data collected, observed retrospectively during 1 year [yr.])
Population: as for outcome 19
Measure: Median (Standard Error); unit: months
Arm/Group | Long Responders to Axitinib
Number analyzed (Participants) | 91
months | 18.727 (2.598)

21. Secondary Outcome: Overall Survival (OS) From Axitinib Treatment in Group of Long Responders
Description: OS was defined as the time from the date of start of axitinib treatment to the date of death due to any cause. If there was no death, the case was censored as OS at latest follow-up.
Time Frame: Day 1 of axitinib dose to death due to any cause or date of latest follow-up in case of censored up to a maximum axitinib therapy of 5.4 years, approximately (from the data collected and observed retrospectively during 1 year)
Population: as for outcome 19
Measure: Median (Standard Error); unit: months
Arm/Group | Long Responders to Axitinib
Number analyzed (Participants) | 91
months | 35.975 (3.453)

22. Secondary Outcome: Number of Participants With Best Response to Axitinib as Second Line of Treatment and Subsequent Treatment in Group of Long Responders
Description: In this outcome measure, data for number of participants with best response to axitinib as second line of treatment and subsequent treatment was collected. Best response is CR and PR, SD or PD. As per RECIST1.1 criteria: CR = disappearance of all target lesions; PR = >= 30% decrease in sum of target lesions taking as reference baseline sum diameters; PD: >= 20% increase in sum of diameters of target lesions, taking as a reference smallest sum on treatment, the sum must also demonstrate an absolute increase of at least 5 mm, or the appearance of >=1 new lesions; SD =neither shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference smallest sum of diameters while on treatment. Subsequent treatment referred to further treatment after second line of treatment.
Time Frame: From first dose of axitinib as second line of treatment and from first dose of axitinib as subsequent treatment up to a maximum axitinib therapy duration of 5.4 years approximately (data collected and observed retrospectively for 1 year)
Population: FAS population was analyzed. This outcome measure as per protocol was intended to be analyzed only in long responders group.
Measure: Count of Participants; unit: Participants
Arm/Group | Long Responders to Axitinib
Number analyzed (Participants) | 91
Participants
  Axitinib as second line of treatment: number analyzed (Participants) | 59
  Axitinib as second line of treatment: CR+PR | 25
  Axitinib as second line of treatment: SD | 32
  Axitinib as second line of treatment: PD | 0
  Axitinib as second line of treatment: No data | 2
  Axitinib as subsequent treatment: number analyzed (Participants) | 32
  Axitinib as subsequent treatment: CR+PR | 15
  Axitinib as subsequent treatment: SD | 16
  Axitinib as subsequent treatment: PD | 0
  Axitinib as subsequent treatment: No data | 1

23. Secondary Outcome: Progression-free Survival (PFS) to Axitinib as Second Line of Treatment and Subsequent Treatment in Group of Long Responders
Description: PFS was defined as the time from the start of axitinib as second line of treatment and subsequent treatment to disease progression or death by any cause. If there was no progression or death, the case was censored as PFS at date of latest follow-up. As per RECIST 1.1, PD: >= 20% increase in sum of diameters of target lesions, taking as a reference smallest sum on treatment, the sum must also demonstrate an absolute increase of at least 5 mm, or the appearance of >=1 new lesions.
Time Frame: From first dose of axitinib as second line and from first dose of axitinib as subsequent lines to PD/death by any cause/date of latest follow-up if censored up to a max. axitinib therapy of 5.4 yrs. approx. (data collected, observed retrospectively 1 yr.)
Population: as for outcome 19
Measure: Median (Standard Error); unit: months
Arm/Group | Long Responders to Axitinib
Number analyzed (Participants) | 91
months
  Axitinib as second line of treatment: number analyzed (Participants) | 59
  Axitinib as second line of treatment | 18.661 (2.917)
  Axitinib as subsequent treatment: number analyzed (Participants) | 32
  Axitinib as subsequent treatment | 16.559 (1.698)

24. Secondary Outcome: Objective Response Rate (ORR) to Axitinib as Second Line of Treatment and Subsequent Treatment in Group of Long Responders
Description: ORR was defined as the number of participants with CR or PR. As per RECIST1.1 criteria: CR = disappearance of all target lesions; PR = >= 30% decrease in sum of target lesions taking as reference baseline sum diameters.
Time Frame: as for outcome 22
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Long Responders to Axitinib
Number analyzed (Participants) | 91
Participants
  Axitinib as second line of treatment: number analyzed (Participants) | 59
  Axitinib as second line of treatment | 25
  Axitinib as subsequent treatment: number analyzed (Participants) | 32
  Axitinib as subsequent treatment | 15

25. Secondary Outcome: Clinical Benefit Rate (CBR) to Axitinib as the Second Line of Treatment and Subsequent Treatment in Group of Long Responders
Description: CBR was defined as the frequency of participants with CR, PR or SD. As per RECIST1.1 criteria: CR = disappearance of all target lesions; PR = >= 30% decrease in sum of target lesions taking as reference baseline sum diameters; PD: >= 20% increase in sum of diameters of target lesions, taking as a reference smallest sum on treatment, the sum must also demonstrate an absolute increase of at least 5 mm, or the appearance of >=1 new lesions; SD =neither shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference smallest sum of diameters while on treatment.
Time Frame: as for outcome 22
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Long Responders to Axitinib
Number analyzed (Participants) | 91
Participants
  Axitinib as second line of treatment: number analyzed (Participants) | 59
  Axitinib as second line of treatment | 57
  Axitinib as subsequent treatment: number analyzed (Participants) | 32
  Axitinib as subsequent treatment | 31

26. Secondary Outcome: Time to Progression (TTP) to Axitinib as the Second Line of Treatment and Subsequent Treatment in Group of Long Responders
Description: TTP was defined as the time from the start of second line of treatment and subsequent treatment to date of disease progression. If there was no progression, the case was censored as TTP at latest follow-up. PD: >=20% increase in sum of diameters of target lesions, taking as a reference smallest sum on treatment, the sum must also demonstrate an absolute increase of at least 5 mm, or the appearance of >=1 new lesions.
Time Frame: From first dose of axitinib as second line of treatment and from first dose of axitinib as subsequent treatment to PD/date of latest follow-up if censored up to max. treatment duration of 5.4 yrs., approx. (data collected, observed retrospectively 1 year)
Population: as for outcome 19
Measure: Median (Standard Error); unit: months
Arm/Group | Long Responders to Axitinib
Number analyzed (Participants) | 91
months
  Axitinib as second line of treatment: number analyzed (Participants) | 59
  Axitinib as second line of treatment | 21.388 (4.695)
  Axitinib as subsequent treatment: number analyzed (Participants) | 32
  Axitinib as subsequent treatment | 18.136 (3.857)

27. Secondary Outcome: Overall Survival (OS) to Axitinib as the Second Line of Treatment and Subsequent Treatment in Group of Long Responders
Description: OS was defined as the time from the date of start of second line of treatment and subsequent treatment till the date of death due to any cause. If there was no death, the case was censored as OS at latest follow-up.
Time Frame: From first dose of axitinib as second line of treatment and from first dose of axitinib as subsequent treatment to death due to any cause/date of latest follow-up if censored upto max. of 5.4 yrs., approx. (data collected, observed retrospectively 1 year)
Population: as for outcome 19
Measure: Median (Standard Error); unit: months
Arm/Group | Long Responders to Axitinib
Number analyzed (Participants) | 91
months
  Axitinib as second line of treatment: number analyzed (Participants) | 59
  Axitinib as second line of treatment | 44.813 (10.540)
  Axitinib as subsequent treatment: number analyzed (Participants) | 32
  Axitinib as subsequent treatment | 26.513 (2.925)

28. Secondary Outcome: Duration of Axitinib Treatment: All Participants
Description: Duration of treatment with axitinib was the time from date of start of axitinib treatment to date of end of axitinib treatment or of latest follow-up if not suspended.
Time Frame: Day 1 of axitinib treatment to end of treatment or date of latest follow-up if not suspended for maximum axitinib therapy duration of 5.4 years, approximately (from data collected and observed retrospectively for 1 year)
Population: FAS included all evaluable participants, i.e. all participants who met all the inclusion criteria and none of the exclusion criteria and have received at least 1 dose of axitinib prior to inclusion in the study. As per protocol, no comparison was planned between long responders and refractory participants.
Measure: Median (Full Range); unit: months
Arm/Group | Axitinib (INLYTA)
Number analyzed (Participants) | 157
months | 10.7 [0.7 to 64.9]

29. Secondary Outcome: Percentage of Participants With Titrated (Increased) Doses of Axitinib of More Than 5 Milligram (mg) Twice Daily: All Participants
Description: Percentage of participants whose axitinib dose was titrated and increased to more than 5mg dose at least 1 time in 12 hours (twice daily), are reported in this outcome measure.
Time Frame: For maximum axitinib treatment duration of 5.4 years, approximately (from data collected and observed retrospectively for 1 year)
Population: FAS population was analyzed. Here, "Overall Number of Participants" signifies participants evaluable for this outcome measure. As per protocol, no comparison was planned between long responders and refractory participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Axitinib (INLYTA)
Number analyzed (Participants) | 70
Percentage of participants | 27.1

30. Secondary Outcome: Percentage of Participants With Reduced Doses of Axitinib of More Than 5 Milligram (mg) Twice Daily: All Participants
Description: Percentage of participants whose axitinib dose was reduced 5 mg dose at least 1 time in 12 hours (twice daily) are reported in this outcome measure.
Time Frame: For maximum axitinib treatment duration of 5.4 years, approximately (data collected and observed retrospectively for 1 year)
Population: as for outcome 29
Measure: Number; unit: Percentage of participants
Arm/Group | Axitinib (INLYTA)
Number analyzed (Participants) | 70
Percentage of participants | 72.9

31. Secondary Outcome: Number of Participants With Adverse Events (AE): All Participants
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. Serious adverse events (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; medically important events. AEs included both SAEs and non-SAEs.
Time Frame: For first line treatment: maximum of 6.6 years approximately; for axitinib treatment: maximum of 5.4 years approximately; for post-axitinib subsequent treatments: maximum of 2.9 years approximately (data collected and observed retrospectively for 1 year)
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib (INLYTA)
Number analyzed (Participants) | 157
Participants | 116

32. Secondary Outcome: Number of Participants Receiving Subsequent Treatment Post Axitinib Treatment: All Participants
Time Frame: Upon initiation of subsequent treatment (post axitinib treatment) to a maximum subsequent treatment duration of 2.9 years approximately (from data collected and observed retrospectively for 1 year)
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib (INLYTA)
Number analyzed (Participants) | 138
Participants | 94

33. Secondary Outcome: Number of Participants as Per Number of Subsequent Lines of Treatment Received Post Axitinib Treatment: All Participants
Time Frame: as for outcome 32
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib (INLYTA)
Number analyzed (Participants) | 94
Participants
  1 treatment line | 94
  2 treatment line | 12
  3 treatment line | 7
  4 treatment line | 4

34. Secondary Outcome: Duration of Subsequent Treatments Post Axitinib Treatment: All Participants
Time Frame: as for outcome 32
Population: as for outcome 29
Measure: Median (Full Range); unit: months
Arm/Group | Axitinib (INLYTA)
Number analyzed (Participants) | 93
months | 4.5 [0.0 to 34.3]

35. Secondary Outcome: Number of Participants With First Best Response to Subsequent Treatments Post Axitinib Treatment
Description: Best response is CR and PR, SD or PD. As per RECIST1.1 criteria: CR = disappearance of all target lesions; PR = >= 30% decrease in sum of target lesions taking as reference baseline sum diameters; PD: >= 20% increase in sum of diameters of target lesions, taking as a reference smallest sum on treatment, the sum must also demonstrate an absolute increase of at least 5 mm, or the appearance of >=1 new lesions; SD =neither shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference smallest sum of diameters while on treatment.
Time Frame: From initiation of subsequent treatment (post axitinib treatment) to a maximum subsequent treatment duration of 2.9 years approximately (from data collected and observed retrospectively for 1 year)
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib (INLYTA)
Number analyzed (Participants) | 94
Participants
  PR+CR | 12
  SD | 35
  PD | 33
  Missing data | 14

36. Secondary Outcome: Number of Participants With Reasons to Discontinue Subsequent Treatments Post Axitinib Treatment: All Participants
Description: In this outcome measure, participants who stopped subsequent treatments after axitinib discontinuation due to any reasons like PD, toxicity and others are reported.
Time Frame: as for outcome 35
Population: FAS population was analyzed. This outcome measure as per protocol was intended to be analyzed only in long responders group. Here, "Overall Number of Participants" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib (INLYTA)
Number analyzed (Participants) | 80
Participants
  PD | 60
  Toxicity | 9
  Other | 9
  No data | 2

37. Secondary Outcome: Overall Survival (OS) From Subsequent Treatments Post Axitinib Treatment
Description: OS was defined as the time from the date of randomization to treatment up to the date of death due to any cause.
Time Frame: as for outcome 35
Population: as for outcome 36
Measure: Median (Standard Error); unit: months
Arm/Group | Axitinib (INLYTA)
Number analyzed (Participants) | 94
months | 24.706 (1.396)

ADVERSE EVENTS:
Time Frame: For first line treatment: maximum of 6.6 years approximately; for axitinib treatment: maximum of 5.4 years approximately; for post-axitinib subsequent treatments: maximum of 2.9 years approximately (data collected and observed retrospectively for 1 year)
Description: Same event may appear as AE and SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event.
Arm/Group | Axitinib (INLYTA)
All-Cause Mortality (participants affected / at risk) | 2/157
Serious Adverse Events (participants affected / at risk) | 15/157
Other Adverse Events (participants affected / at risk) | 116/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib (INLYTA) (N=157)
Anemia (Blood and lymphatic system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Pancreatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Pyrexia (General disorders) | 1
Abdominal sepsis (Infections and infestations) | 1
Biliary sepsis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1
Confusional state (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib (INLYTA) (N=157)
Anemia (Blood and lymphatic system disorders) | 6
Polycythaemia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 23
Eyelid oedema (Eye disorders) | 2
Diarrhea (Gastrointestinal disorders) | 76
Nausea (Gastrointestinal disorders) | 17
Vomiting (Gastrointestinal disorders) | 11
Dysgeusia (Gastrointestinal disorders) | 5
Dysphagia (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Pancreatitis (Gastrointestinal disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Ageusia (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 1
Glossodynia (Gastrointestinal disorders) | 1
Odynophagia (Gastrointestinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Hypertension (Vascular disorders) | 40
Asthenia (General disorders) | 66
Hypotension (Vascular disorders) | 2
Pulmonary embolism (Vascular disorders) | 1
Mucosal inflammation (General disorders) | 21
Capillary fragility (Vascular disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 25
Oedema peripheral (General disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 4
Dermal cyst (Skin and subcutaneous tissue disorders) | 1
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1
Pruritus genital (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Pyrexia (General disorders) | 2
Pain (General disorders) | 2
Chest pain (General disorders) | 1
Fatigue (General disorders) | 1
Feeling cold (General disorders) | 1
Hyperhidrosis (General disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 28
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Aphonia (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Gastroenteritis (Infections and infestations) | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Mastitis (Infections and infestations) | 1
Pharyngotonsillitis (Infections and infestations) | 1
Gynaecomastia (Reproductive system and breast disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Fall (Injury, poisoning and procedural complications) | 1
Haematuria (Renal and urinary disorders) | 1
Blood creatinine increased (Investigations) | 14
Hydronephrosis (Renal and urinary disorders) | 1
Oliguria (Renal and urinary disorders) | 1
Alanine aminotransferase increased (Investigations) | 6
Polyuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Insomnia (Psychiatric disorders) | 3
Weight decreased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Paraesthesia (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 2
Haemoglobin increased (Investigations) | 2
Bradyphrenia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Blood triglycerides increased (Investigations) | 1
Paresis (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 21
Hypercalcaemia (Metabolism and nutrition disorders) | 7
Gout (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1

LIMITATIONS AND CAVEATS:
Prioritization of outcome measures was based on sponsor's discretion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT03538717/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT03538717/SAP_001.pdf